CLINICAL TRIAL: NCT04392115
Title: PRomoting Exercise During the Pandemic to Increase Activity and Reduce Effects of Social Isolation for COVID: The PREPARE for COVID Trial
Brief Title: The PREPARE for COVID Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Record Dates: First submitted 2020-05-15; First posted 2020-05-18 (Actual); Last update posted 2020-05-18 (Actual); Status verified 2020-05

CONDITIONS: Comorbidities and Coexisting Conditions; Social Isolation
Keywords: COVID-19; Virtual care; Older adults; Exercise; Social Isolation
MeSH Terms: conditions — Social Isolation; COVID-19; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Experimental): The home-based exercise program called the PREPARE program.
  Exercise will be prescribed as one-hour sessions, performed a minimum of three times per week for at least three months, consisting of: 1) strength training; 2) aerobic exercise and 3) flexibility.
  Interventions: Behavioral: The PREPARE program
- Control Group (No Intervention): The control group will receive the World Health Organization recommendations for physical activity for people greater or equal to the age of 65 years old pamphlet, as well as a guide to healthy eating for older adults.

INTERVENTIONS:
Behavioral: The PREPARE program — A home-based exercise program guided by paper materials, weekly phone calls, and a DVD.
  Exercise will be prescribed as one-hour sessions, performed a minimum of three times per week for at least three months, consisting of: 1) strength training; 2) aerobic exercise and 3) flexibility.
  Arms: Exercise Group

SUMMARY:
This is a randomized trial of home-based exercises versus control for older adults during the COVID-19 pandemic. The hypothesis is that participation in a home-based program will reduce the risk of adverse effects of physical distancing by decreasing patient-reported disability, improving mental health and avoiding hospitalization or institutionalization for vulnerable older people

DETAILED DESCRIPTION:
Background:More than 6.5 million Canadians are > 65 years of age. Over half of older Canadians live with multiple comorbidities, leaving them at high risk of adverse outcomes of COVID-19. Social isolation and physical distancing orders are especially important to protect the health of this high-risk population. Vulnerable older Canadians are also at high risk of physical and mental health deterioration caused by the physical distancing meant to protect them from COVID-19. Effective management of the COVID-19 pandemic and its consequences will require evidence-based strategies to support isolated vulnerable older Canadians. Exercise interventions can reduce the adverse health effects of social isolation and demonstrate larger effect sizes in older people with comorbidities. However, no exercise interventions have been tested in an acute isolation scenario such as the COVID-19 pandemic, which also requires that exercise interventions be home-based and remotely supported, presenting unique challenges to participation and adherence.

Our team is uniquely positioned re-orient proven and robust programming, supported by a national network of investigators and existing infrastructure. We can immediately launch a large-scale trial to test the effectiveness of a remotely supported home exercise program (designed in partnership with vulnerable older Canadians) to mitigate the negative consequences of physical distancing to keep older Canadians healthy and safe from COVID-19. We hypothesize that participation in the PREPARE program will decrease the individual, health system and population health impacts of COVID19 induced physical distancing and social isolation.

Research aims:Estimate the effectiveness of a remotely supported, home-based multimodal exercise program for older people with multiple comorbidities to improve our primary outcome: patient-reported disability 90-days after enrollment; secondary outcomes: patient-centered (depression, anxiety, quality of life, frailty, survival, 1-year disability scores, COVID19 severity) and system-relevant (admissions, emergency visits, institutionalization, costs, cost-effectiveness).

Methods: Design, setting and participants: Parallel-arm multicenter randomized controlled trial at 3 Canadian hospitals. People >65 years old recently discharged home with >2 comorbidities will be included. Intervention: Three month supported home-based exercise program with demonstrated efficacy, feasibility and acceptability for vulnerable older people.

Outcomes and sample size: We will have 90% power to detect a clinically important difference of in our primary outcome (validated WHODAS tool, 90-days post-enrollment) with 372 participants (186/arm)

ELIGIBILITY:
Inclusion Criteria:

* 65 years of age or older
* 2 or more co-morbidities
* recent discharge from hospital

Exclusion Criteria:

* Inability to communicate in English or in French
* Unreachable by telephone
* Unstable cardiovascular or valvular disease
* Discharged to Long-Term Care

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 372 (Estimated)
Dates: Start 2020-06-15 (Estimated); Primary Completion 2020-12-15 (Estimated); Study Completion 2021-09-15 (Estimated)

PRIMARY OUTCOMES:
Patient-reported disability 90 days after enrollment | Assessing change in score from baseline data collection to 90 days from enrollment
  The World Health Organization Disability Assessment Schedule 2.0 (WHODAS) will be used . It is a patient-reported disability scale that assesses limitations in six major life domains - cognition, mobility, self-care, social interaction, life activities and participation in society. Participants will report if they have had no difficulty, mild difficulty, moderate difficulty, severe difficulty or extreme difficulty (simply cannot do) with the items listed.

SECONDARY OUTCOMES:
Mental Health | Assessing change in the participants GAD-7 score from baseline to monthly scores for 12 months.
  The Patient Health Questionnaire-9 item (PHQ-9) and the Generalized Anxiety Disorder 7-item (GAD-7) are validated tools for diagnosing anxiety and depression.
Function | Monthly step count from enrollment to monthly step counts for 12 months from enrollment.
  Step count using pedometer
Health-related quality of life | Assessing change in the participants EQ-5D-5L score from baseline to monthly scores for 12 months.
  The EQ-5D-5L is a validated instrument with Canadian valuation statistics and national use, which informs incremental cost per quality-adjusted life year gained.
Frailty | Assessing change in the participants CFS score from baseline to monthly scores for 12 months.
  The Clinical Frailty Scale (CFS) provides a global assessment of frailty.
All-cause mortality. | From enrollment to 12 months after enrollment.
  All deaths and death dates will be identified via chart review or telephone call.
Health System - Emergency Department Visits | Monthly for 12 months following enrollment.
Health System - Re-admission | Monthly for 12 months following enrollment.
Health System - Transfer to Long-Term Care | Monthly for 12 months following enrollment.
COVID-19 test results | Monthly for 12 months following enrollment.
Safety [Adverse Events] | Assessing frequency of, or change in any safety events from enrollment up to 90 days from enrollment between the exercise group and control group.
  Falls, cardiac or respiratory complications and unplanned healthcare encounters will be collected during the exercise treatment period for the exercise group. For the control group, participants will be asked if they experienced any falls since the time of enrollment up until the day before surgery. Unplanned healthcare encounters will also be collected during the time of enrollment to the final day of the exercise intervention for the intervention group through chart review.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel I McIsaac, MD, Principal Investigator — The Ottawa Hospital Research Institute